## STATISTICAL ANALYSIS PLAN For

## An Open-Label Phase 2a Study to Evaluate the Safety and Efficacy of AVB-S6-500 in Patients with IgA Nephropathy

## PROTOCOL NUMBER: AVB500-IGA-001 NCT04042623

Sponsor:

Aravive, Inc

3730 Kirby Drive, Ste 1200

Houston, Texas 77098

**USA** 

Document Date:

20 October 2021

Aravive, Inc. certifies that Statistical Analysis Plan was not drafted, since the study was terminated after only one patient was enrolled in the study AVB500-IGA-001. This subject received a single dose of the study drug and did not complete the study. No outcome measures were analyzed and there are no plans to conducted any analyses in the future.

Confidential Page 1 20 October 2021